CLINICAL TRIAL: NCT02047292
Title: Dynamic Range of Motion (ROM) Assessment Using Gait Analysis and Three-dimensional Fluoroscopy in Patients Treated by Total Hip Arthroplasty (THA) With Different Head Diameters
Brief Title: Dynamic ROM Via Gait Analysis and 3D Fluoroscopy in THA With Different Head Diameters
Acronym: DROMDP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: DePuy International (Industry)
Responsible Party: Principal Investigator, Alberto Leardini, DPhil, Alberto Leardini, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IORDePuyD57613
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Hip Osteoarthritis
Keywords: Gait analysis; 3D videofluoroscopy; Femoroacetabular impingement; Neck-cup impingement; Head-neck ratio; Hip scores; Functional assessment; Cup size; Range of motion; Unilateral Primary; Secondary
MeSH Terms: conditions — Osteoarthritis, Hip; Femoracetabular Impingement; Neoplasm Metastasis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- THA28 (Active Comparator): THA Corail PinnacleCoC28
  Interventions: Device: THA Corail PinnacleCoC28
- THA36 (Active Comparator): THA Corail DeltaMotion36
  Interventions: Device: THA Corail DeltaMotion36
- THA40 (Active Comparator): THA Corail DeltaMotion40
  Interventions: Device: THA Corail DeltaMotion40

INTERVENTIONS:
Device: THA Corail PinnacleCoC28 — Uncemented THA with Corail stem and Pinnacle acetabular cup with CoC 28 mm head
  Arms: THA28
Device: THA Corail DeltaMotion36 — Uncemented THA with Corail stem and DeltaMotion acetabular cup with 36 mm head
  Arms: THA36
Device: THA Corail DeltaMotion40 — Uncemented THA with Corail stem and DeltaMotion acetabular cup with 40 mm head
  Arms: THA40

SUMMARY:
Pain and reduced function are the most common symptoms of coxarthritis. Pain relief and normal range of motion (ROM) restoration are the objectives of a Total Hip Arthroplasty (THA) procedure. It is recognized that increased head-neck ratio results in increased ROM due to the fact that prosthetic impingement between neck and acetabular liner occurs with wider arcs of motion. This head-neck ratio has been investigated extensively only in vitro (on cadavers or sawbones) or using mathematical modeling in computer simulations. These studies are limited by the lack of soft tissues and muscle activations in the models. This study will clinically assess the effect of prosthetic head diameter on patient capability of performing movements which require extreme arcs of motion of the hip joint. Therefore, the research questions are:

* What role do soft tissues play in limiting ROM?
* Can prosthetic impingement really occur in a well positioned THA?
* Can a bigger head diameter alone reduce the risk of impingement?

DETAILED DESCRIPTION:
This will be a prospective comparative randomized double-blind Study (both patient and the clinical engineer performing the gait analysis will be blind with respect to the prosthetic head diameter implanted). Patient recruitment will last 12 months and the Study will have a follow-up period of 12 months. A total number of 45 patients will be recruited. Patients will be randomly allocated into three groups: the first group will undergo THA with a 28mm diameter head (Pinnacle Acetabular System, with a ceramic on ceramic - CoC - bearing), in the second group THA will be performed using a 36 mm diameter head (DeltaMotion), finally patients in the third group will undergo THA with a 40 mm diameter head (DeltaMotion). Patients will be operated by three surgeons of the same hospital according to the same surgical procedure and using the same direct lateral approach. All patients will receive a Corail stem and will follow the same rehabilitation program.

* Primary endpoint: Gait analysis and fluoroscopy will provide quantitative information of prosthesis in vivo performance, e.g. what is the arc (degrees) of active or passive motion when prosthetic impingement occurs?
* Secondary endpoint(s): these analyses will also allow to: 1) assess ROM of the operated hip versus contralateral non operated hip and the effect of prosthetic head diameter and any correlation to hip functional scores validated and commonly used in the Literature; 2) set reproducible criteria for in vivo fluoroscopic analysis of ROM in THA patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with unilateral primary or secondary hip arthrosis indicated for THA;
* Men and female, age between 35 and 55 years old;
* BMI smaller than 30;
* Patients able to understand the protocol and to sign the informed consent.

Exclusion Criteria:

* Child-bearing female;
* Patients with also controlateral hip arthritis;
* Neurological patients, because of possible alteration of neuro-muscular control of the replaced hip;
* Patients treated with joint replacement at any other lower limb articulation

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
Number of Participants and Hip Joint Positions with the Occurrence of Implant Impingement | 12 months
  Three-dimension videofluoroscopy is used to calculate prosthesis component relative pose, and to estimate minimum distance at the areas of risk of impingement
Number of Participants with Functional Deficits at the Hip Joint as Measured by Gait Analysis | 12 months
  Three-dimension kinematics and kinetics of the trunk, pelvis and lower limb joints is used during level walking and other motor tasks, as well as for the single exercises of hip joint extreme motion analyzed in videofluoroscopy, to assess thoroughly those patients with and without impingement.

SECONDARY OUTCOMES:
Range of Motion of the operated hip versus contralateral non-operated hip | 12 months
  Standard clinical range of motion at the two hips
Correlations between prosthetic head diameter and hip functional scores | 12 months
  The effect of prosthetic head diameter and any correlation to hip functional scores validated and commonly used in the Literature
Standard Clinical Hip Scores | pre-op, and 12 months
  Outcomes: Harris Hip Score, Oxford Hip Score, WOMAC, Forgotten Joint score and UCLA activity score will be assessed and recorded pre-operatively and post-operatively at one year after surgery.
X-ray measurements | 12 months
  Radiographic assessment will also be performed at one year after surgery to assess implant position and osteointegration

CONTACTS AND LOCATIONS:
Overall Officials: Sandro Giannini, MD, Prof, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, BO, Italy

REFERENCES:
- See also: Istituto Ortopedico Rizzoli — http://www.ior.it/